CLINICAL TRIAL: NCT02257411
Title: A Simple Method to Determine the Size of the ProSeal LMA (PLMA) in Children
Brief Title: A Method to Determine the Size of Laryngeal Mask Airway (LMA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University Hospital (Other)
Responsible Party: Principal Investigator, Murat Haliloglu, Medical doctor, Yeditepe University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Triple
Other Study IDs: 346
Record Dates: First submitted 2014-09-22; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Ear Based ProSeal LMA
Keywords: child; ear based; Proseal LMA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ear-sized based and weight based formula (Active Comparator): the sizes of the PLMA determined with the ear-based compared with the sizes according to the manufacturer's weight-based formula
  Interventions: Device: Ear-sized based

INTERVENTIONS:
Device: Ear-sized based — the sizes of the PLMA determined with the ear-based formula were compared with the sizes according to the manufacturer's weight-based formula

SUMMARY:
After institutional ethics board approval and written informed consent from parents, 197 children scheduled for routine genitourinary operation and in whom a LMA was indicated for anesthesia were included in the study. The size of the LMA was determined by choosing the size that was best matched with the auricle of the children. The results were compared with the standard method recommended by the manufacturer's weight-related guidelines. The patients were classified in different groups depending on the PLMA sizes determined by both methods. A kappa coefficient evaluated the agreement between both techniques.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I/II
* scheduled for genitourinary operation
* LMA was indicated for anesthesia

Exclusion Criteria:

* surgery lasting more than 3 h
* overweight or underweight patients
* gastroesophageal reflux
* risk of aspiration
* airway infection in the last six weeks
* decreased pulmonary or chest wall compliance.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 197 (Actual)
Dates: Start 2013-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
the sizes of the PLMA determined with the ear-based formula | One year
  we were to determine whether the size of the auricle could be used as a proxy for the appropriate size of the PLMA

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University Hospital, Istanbul, Kozyatağı, Turkey (Türkiye)